CLINICAL TRIAL: NCT04690998
Title: Outcome Measures and Biomarkers in a Cohort of Spinal Muscular Atrophy Type III/ IV Patients
Acronym: SMOB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-54
Record Dates: First submitted 2020-10-20; First posted 2020-12-31 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without treatment for SMA (Other): Patient that will not take treatment for SMA during the two years of the study.
  Interventions: Other: Blood Samples; Other: MRI
- Under treatment for SMA (Other): Patient that will take treatment for SMA during the two years of the study
  Interventions: Other: Blood Samples; Other: MRI

INTERVENTIONS:
Other: Blood Samples — Genetic, proteomic, neurofilament analysis
Other: MRI — Spinal and muscular MRI

SUMMARY:
The "SMOB" project intends to contribute to fill the gap with reliable and operational outcome measures for type III and IV SMA. In analysing the reliability in imaging (spinal and muscular), electrophysiology analysis (MUNIX), and evaluate the evolution of respiratory function for 50 patients' cohort. The investigators would also take the opportunity to collect biologic samples in order to investigate genetic markers and to assess quality of life of patients by QoL-gNMD questionnaire. The investigators aim to build a database that will allow us to evaluate the effectiveness of a new therapy for adult SMA patients by studying the natural history of the disease. The investigators have distributed the various expertise in Work Package where several centers are involved.

This study is original in that it evaluates the parameters of qMRI and MUNIX in correlation with blood biomarkers. To our knowledge, there are no quantitative MRI (spinal and muscular) biomarkers and/or electrophysiological (MUNIX technique) highlighted for tracking the progression of the adult form of SMA type III and IV. This pilot study would allow identification of predictive markers of the disease progression, and to have validated, sensitive to change and relevant measurement tools that could be used as endpoints in future therapeutic trials.

DETAILED DESCRIPTION:
Spinal muscular atrophy is an autosomal recessive neurodegenerative disease characterized by degeneration of spinal cord motor neurons, atrophy of skeletal muscles, and generalized weakness. It is caused by homozygous disruption of the survival motor neuron 1 (SMN1) gene by deletion, conversion, or mutation. Spinal muscular atrophy (SMA) is a genetic disease that affects mostly children but also some adults. Motor neuron loss often results in severe muscle weakness causing affected infants to die before reaching 2 years of age. There are types I, II, and III that affect children, and Type IV that affects adults. The prevalence of this rare disease is around 1/30 000 births.The disease is characterized by a slowly progressive muscle weakness over many years in patients with a milder form.

SMA is caused by the loss of SMN1 and the retention of at least 1 copy of a highly homologous SMN2. An alternative splicing event in the pre-mRNA arising from SMN2 results in the production of low levels of functional SMN protein. Onset and severity of disease, and therefore type, correlate mainly with SMN2 copy number (and theoretically with SMN protein level) providing a molecular basis for the classification of the different subtypes of SMA. Type III patients have 3-4 copies, and patients with type 4 usually have 4 copies or more. About 30% of patients have type III SMA, which is associated with onset between ages 18 months and adulthood. By definition standing or walking without support is achieved, although many patients lose these abilities later with disease progression (Zerres.K et al 1995). Patients usually present with symptoms of falls, difficulty climbing stairs, and other features of proximal weakness and respiratory deficit. Abnormal gait characteristics are common in order to compensate for weakness, and many patients are able to continue ambulation despite severe weakness. Foot deformity may be seen in ambulatory patients. Lifespan is normal in SMA type III. Some classifications of SMA include an additional disease subtype at the mild end of the continuum. In this case, patients may be classified as having type IV SMA. Patients with type IV, representing less than 5% of SMA, are ambulatory and have the mildest form of SMA. The presentation is very similar to type III and is distinguished solely on later onset during adulthood (Zerres K. et al 1995, Piepers S. et al 2008). Though onset of type IV is not clearly defined, it is often considered to be at age 30 or later. The remarkably slow rate of progression of late onset SMA types IIIb and IV underlines that more sensitive tools are needed to monitor muscle strength in clinical trials.

Documenting functional status in SMA is important, since all patients show limitations in daily functioning and the preservation or improvement is the goal for pharmacological intervention. Regardless, precisely designed supportive, rehabilitative, and palliative care can partly reduce the disease burden and alter the natural history. Treatment is designed to address the primary and secondary effects of muscle weakness and should include management of pulmonary complications, nutritional and gastrointestinal support, orthopedic care, rehabilitative interventions, and end-of-life care. Standards of care for SMA are established, but there is need for improved and more specific directives in this regard (Wang CH et al 2007). It is important to understand the expected natural history of SMA to anticipate and stratify risk, to monitor function with appropriate measures, to determine the appropriate treatment options, and to delivery timely intervention. Proactive care and treatment decision-making by the treatment team and family are of utmost importance. Preclinical progress in the SMA field has been rapid since the identification of SMN1 as the responsible gene in 1995 and by the creation of the first mouse model in 2000 (Hsieh-Li HM et al, 2000).

Several clinical therapeutic trials have been performed in SMA without success. The first very successful therapies in murine models of SMA were published in 2010 using gene therapy to replace the SMN1 gene (Foust KD et al, 2010). Later a phase 1 trial was conducted using systemic delivered AAV9 gene therapy to replace SMN1 in infants with SMA type I. A single intravenous infusion of adeno-associated viral vector containing DNA coding for SMN resulted in longer survival, superior achievement of motor milestones, and better motor function than in historical cohorts (Mendell. R et al, 2017). More recently, development of antisense oligonucleotide therapies that can modify SMN2 splicing to include exon 7 and produce increased amounts of full length SMN protein has shown promising results. Nusinersen is an antisense oligonucleotide. It has been developed for the treatment of spinal muscular atrophy (SMA). In the CHERISH trial, among children with later onset SMA, significant improvement in motor function was observed with Nusinersen treatment as compared with a sham procedure. Persons with later-onset SMA and their caregivers indicated that stabilization of their current state would meet their therapeutic expectations and represent a clinically meaningful response. In this trial, as in the ENDEAR trial for infantile-onset SMA (most likely to be classified as SMA type 1), they found that Nusinersen had the capacity to produce meaningful changes in the clinical course of SMA. In this trial, more than half the children in the Nusinersen group had an increase from baseline to month 15 in the Hammersmith Functional Motor Scale-Expanded (HFMSE) score of at least 3 points (i.e., a clinically meaningful improvement), which is uncommon among children with later-onset SMA (Mercuri E. et al, 2018). This trial had some limitations, no adult form of SMA was considered. In the trial, 16% of the enrolled children were 6 years of age or older. The results reported are consistent with the results of previous open-label studies that enrolled children up to 15 years of age. The studies showed that Nusinersen had positive effects in populations of children with SMA type II or III that were broader and more heterogeneous than the population enrolled in this trial. That is why it is important to explore the Nusinersen effects on type III and IV and allow adult patients to benefit from this new therapy. For that it is essential to have efficient biomarkers for evaluation of efficiency of Nusinersen as it remains somewhat controversial given its high price and its highly invasive administration. In this therapeutic evaluation context, the choice of outcome measures had a great importance. Moreover, although advances have been made on SMA pathogenesis, there still are unknown factors that could explain the variability of the disease's severity among patients.

The "NH-SMA" project intends to contribute to fill the gap with reliable and operational outcome measures for type III and IV SMA. In analysing the reliability in imaging (spinal and muscular), electrophysiology analysis (MUNIX), and evaluate the evolution of respiratory function for 50 patients' cohort. The investigators would also take the opportunity to collect biologic samples in order to investigate genetic markers and to assess quality of life of patients by QoL-gNMD questionnaire. The investigators aim to build a database that will allow us to evaluate the effectiveness of a new therapy for adult SMA patients by studying the natural history of the disease. The investigators have distributed the various expertise in Work Package where several centers are involved.

This study is original in that it evaluates the parameters of qMRI and MUNIX in correlation with blood biomarkers. To our knowledge, there are no quantitative MRI (spinal and muscular) biomarkers and/or electrophysiological (MUNIX technique) highlighted for tracking the progression of the adult form of SMA type III and IV. This pilot study would allow identification of predictive markers of the disease progression, and to have validated, sensitive to change and relevant measurement tools that could be used as endpoints in future therapeutic trials.

The primary objective is to identify potential markers (clinical, biological, genetic, imaging) of the health status evolution The health evolution will be assessed at 6, 12, 18 and 24-month post-inclusion. The primary point is the 24-month follow-up. The other points will be retained as secondary points.

The health status evolution will be assessed using

* Clinical examination :
* MFM-32 (gold standard, Motor Function Measure), RULM (Revised Upper Limb Module) HFMSE (Hammersmith Functional Motor Scale Expanded), SMAFRS (spinal muscular atrophy functional rating scale)
* Muscle strength assessment (QMT)
* gait speed, 30s sit to stand, climb 4 stairs
* Evaluation of Respiratory Functions
* Quality of life, pain, and fatigue assessment: QoL-NMD-V1, EVA, EVN, FSS
* Imagery: Muscular, spinal and cranial MRI
* Electrophysiological examination
* Biological and biochemical analyses: blood test samples, NF dosage, genetics, proteomics, biobanking The main analyses currently used to determine the patient status are the clinical examination, especially the MFM-32 score, which is the gold standard, the RULM and the evaluation of the respiratory functions. The other analyses will bring supplementary data. Their comparison to the usual analyses will allow us to see if it is possible to detect more subtle changes in the patient status.

The secondary objectives are to identify potential markers (clinical, biological, genetic, imaging) of the treatment response in the subgroup of patients who will be treated The treatment response will be assessed at 6, 12, 18 and 24- month post-inclusion.

The treatment response will be assessed This study is a multicenter, prospective study, to follow for 24 months a cohort of 100 patients aged from 18 to 70 and suffering from type III and IV SMA.

The choice of a prospective study is most likely to fulfill the objectives. Five evaluation visits are planned at D0, M6, M12, M18 and M24. Two years follow-up is necessary because of the variability and the rate of progression of this chronic disease. This period is also appropriated to better estimate the clinically meaningful difference of the outcome measures studied. Thus, a 24 month- follow-up will be conducted with a visit every one year. An inter-visit questionnaire will be completed by phone once a year between 2 visits, to have a more regular follow-up of the disease evolution and to minimize the number of patients lost to follow-up.

100 patients will be included. The investigators estimate than 70 will be able to walk independently and 30 in wheelchairs. About 40 type III patients will be treated with Nusinersen during the 2 years follow-up and won't be evaluated for natural history of SMA.

The sample size will allow to approximate pertinent odd ratios regarding the primary (health status evolution) and the secondary (treatment response) objectives.

The study will assess markers of 1) health status evolution; 2) treatment response.

The health status evolution will be assessed at 6, 12, 18, and 24-month post-inclusion. The health status will be measured from many parameters (Clinical examination, Imagery, Electrophysiological examination Biological and biochemical analyses) The treatment response will be assessed in the subgroup of treated patients, at 6- 12- 18- and 24-month post-inclusion. The response treatment will be assessed through the improvement of clinical scores, and quality of life Predictive biomarkers of disease progression of type III and IV SMA will be evaluated from the baseline to the end of the study

It is expected that this study will help to identify quantitative reliable markers that will allow a better understanding of the disease progression and a better management and patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Between 18 and 70 years old
* Given written informed consent after being informed of the purpose, progress and potential risks

Exclusion Criteria:

* Concomitant impairment of central nervous system (for example cervical myelopathy)
* Homeless patients
* Deprived of their liberty by a court or administrative order or under guardianship
* Unable to understand the purpose and conditions of carrying out the study, unable to give consent
* Patients included in another clinical trial or exclusion period from a previous clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Clinical examination | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  MFM-32 Score
VAS | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  Pain, tiredness, depression
Fatigue Severity Scale (FSS) | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  Pain, tiredness, depression
Muscle strength | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  Hand grip , tibialis anterior, forearm and hands circumference, ankle dorsiflexion
Timed test | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  Walk 10 meters
Timed test | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  6 min walk
Timed test | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  30 sit to stand
Pulmonary function test | Change from Baseline at 12 months and 24 months
  FVC, MIP, MEP
Quality of Life of patients | Change from Baseline at 6 months, 12 months, 18 months, 24 months
  QoL-gNMD
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of SMN copy number gene and protein
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of Neurofilament
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of phosphorylated Neurofilament
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of transcriptomics
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of proteomics
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of microRNA, circulatingRNA, DNA methylation, circulating DNA
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of microRNA
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of circulatingRNA
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of DNA methylation, circulating DNA
Blood samples | Change from Baseline at 12 months and 24 months
  Analysis of circulating DNA
MRI | Change from Baseline at 24 months
  Muscular MRI
MRI | Change from Baseline at 24 months
  Spinal MRI

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Service de Neurologie,Hôpital Raymond-Poincaré, Garches
  - Département de Neurologie - CHRU Lille, Lille
  - Service ENMG - Pathologies neuromusculaires, centre de référence en pathologie neuromusculaire Rhône-Alpes, Centre de référence SLA, Lyon
  - CHU Montpellier, Montpellier
  - Service Laboratoire d'Explorations Fonctionnelles, Hôtel-Dieu, CHU Nantes, Nantes
  - Centre de Référence des Maladies Neuromusculaires - Pôle Neurosciences Cliniques, CHU Nice, Nice
  - Institut de Myologie, Paris
  - Service de Neurologie - CHU Saint-Etienne, Saint-Etienne
  - Service des Maladies Neurologiques Rares, Saint-Pierre
  - Centre de référence des Maladies Neuromusculaires,Service de Neurologie, Hôpital de Hautepierre, Strasbourg
  - Service de Neurologie et d'explorations fonctionnelles, Hôpital Pierre-Paul Riquet, Place du Docteur Baylac, Toulouse

IPD SHARING:
Plan to Share IPD: No